CLINICAL TRIAL: NCT05478603
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL GROUP STUDY TO COMPARE THE PHARMACOKINETICS OF PF-07081532 IN ADULT PARTICIPANTS WITH VARYING DEGREES OF HEPATIC IMPAIRMENT RELATIVE TO PARTICIPANTS WITHOUT HEPATIC IMPAIRMENT
Brief Title: A Study to Understand How the Study Medicine (PF-07081532) is Processed in People With Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C3991009
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-04

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Hepatic impairment; Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: PF-07081532 Participants without hepatic impairment (Experimental): Participants without hepatic impairment will receive a single 20 mg dose of PF-07081532, administered orally as 1 PF-07081532 20 mg tablet.
  Interventions: Drug: PF-07081532
- Group 2: PF-07081532 Participants with mild hepatic impairment (Experimental): Participants with mild hepatic impairment will receive a single 20 mg dose of PF-07081532, administered orally as 1 PF-07081532 20 mg tablet
  Interventions: Drug: PF-07081532
- Group 3: PF-07081532 Participants with moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment will receive a single 20 mg dose of PF-07081532, administered orally as 1 PF-07081532 20 mg tablet.
  Interventions: Drug: PF-07081532
- Group 4: PF-07081532 Participants with severe hepatic impairment (Experimental): Participants with severe hepatic impairment will receive a single20 mg dose of PF-07081532, administered orally as 1 PF-07081532 20 mg tablet.
  Interventions: Drug: PF-07081532

INTERVENTIONS:
Drug: PF-07081532 — PF-07081532 20 milligrams (mg), 1 tablet orally, once on Day 1

SUMMARY:
The purpose of this study is to understand the effects of liver functional impairment on the study medicine (PF-07081532). People with liver functional impairment may process the study medicine differently from healthy people.

We are seeking participants who:

* Are between 18 and 70 years of age;
* Have a BMI (body mass index) of 17.5 to 38.0 kg/m2, inclusive, and a total body weight >50 kg (110 lbs.).

Participants will take the study medicine as a tablet once at the study clinic, and then will stay onsite for about 7 days. During this time, the study team will monitor their treatment experience and take some blood samples to test the level of PF-07081532. This will help us understand if certain level of liver functional impairment could affect the study medicine being processed in the body.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 70 years, inclusive at the screening visit.
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* BMI of 17.5 to 38.0 kg/m2, inclusive, and a total body weight >50 kg (110 lb).
* Group 1 only: at screening, no clinically relevant abnormalities identified by a detailed medical history, physical exam, including blood pressure and pulse rate measurement, ECG and clinical laboratory tests.
* Group 1 only: no known or suspected hepatic impairment and meet the criteria based on screening laboratory liver function tests.
* Groups 2, 3 & 4 only: stable hepatic impairment that meets criteria for Class A, B, or C of the Child-Pugh classification with no clinically significant change in disease status within 28 days before screening.
* Groups 2, 3 & 4 only: stable concomitant medications for the management of individual participant's medical history.

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* At screening, a positive result for HIV antibodies.
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2), or participants with suspected MTC per study doctor's judgement.
* History of acute pancreatitis within 6 months before the screening visit or any history of chronic pancreatitis.
* Other medical or psychiatric condition or laboratory abnormality that may increase the risk of study participation or make the participant inappropriate for the study.
* Use of specific prohibited prior/concomitant therapies
* Use of an investigational product within 30 days (or local requirement) or 5 half-lives (whichever longer).
* eGFR<60 mL/min/1.73m2 at screening.
* A positive urine drug test at screening or admission to study clinic.
* At screening or admission to study clinic, a positive breath alcohol test.
* For females, pregnancy, as indicated by a positive serum pregnancy test at screening and/or positive urine pregnancy test in women capable of having children at admission to study clinic
* Group 1 only: evidence of chronic liver disease including history of hepatitis, hepatitis B, or hepatitis C.
* Group 1 only: history of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of screening.
* Group 1 only: screening ECG demonstrating QTcF interval >450 ms or a QRS interval >120 ms.
* Group 1 only: screening seated systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg
* Group 1 only: use of chronic prescription medications within 7 days or 5 half-lives (whichever longer) before Day 1, or for prohibited medications, use within the required washout/restriction period.
* Group 2, 3 & 4 only: Hepatic carcinoma or hepatorenal syndrome or limited predicted life expectancy (defined as <1 year in Groups 2 & 3 and <6 months for Group 4 only).
* Group 2, 3 & 4 only: a diagnosis of hepatic dysfunction secondary to any acute ongoing hepatocellular process that is documented by medical history, physical exam, liver biopsy, hepatic ultrasound, CT scan, or MRI.
* Group 2, 3 & 4 only: history of surgery that would be expected to alter absorption, distribution, metabolism, or excretion properties of PF-07081532.
* Group 2, 3 & 4 only: history of gastrointestinal hemorrhage due to esophageal varices or peptic ulcers less than 4 weeks prior to screening.
* Group 2, 3 & 4 only: signs of clinically active Grade 3 or 4 hepatic encephalopathy
* Groups 2, 3 & 4 only: severe ascites and/or pleural effusion, except for those categorized in Group 4 who may be enrolled provided participant is medically stable, per the study doctor's judgment.
* Groups 2, 3 & 4 only: previously received a kidney, liver, or heart transplant.
* Groups 2, 3, & 4 only: screening ECG demonstrating a QTcF interval >470 ms or a QRS interval >120 ms.
* Groups 2, 3 & 4 only: at screening, admission to study clinic or pre-dose on Day 1, persistent severe, uncontrolled hypertension.
* Groups 2, 3 & 4 only: ALT or AST >5x upper limit of normal on clinical laboratory tests at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991009

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 39 participants were screened, of whom 24 participants were assigned to treatment and treated, with 6 participants in each group (without hepatic impairment, with mild hepatic impairment, with moderate hepatic impairment, and with severe hepatic impairment).
Groups:
- Without Hepatic Impairment: This arm included participants without hepatic impairment who received PF-07081532 20mg on Day 1.
- Mild Hepatic Impairment: This arm included participants with mild hepatic impairment who received PF-07081532 20mg on Day 1.
- Moderate Hepatic Impairment: This arm included participants with moderate hepatic impairment who received PF-07081532 20mg on Day 1.
- Severe Hepatic Impairment: This arm included participants with severe hepatic impairment who received PF-07081532 20mg on Day 1.
Period: Overall Study
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 6 | 6 | 6 | 6
Completed (The entire study including follow-up phase.) | 6 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who each took 1 dose of PF-07081532.
Groups:
- Total: Total of all reporting groups
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 0 | 1 | 1 | 0 | 2
  45-64 years | 6 | 3 | 2 | 5 | 16
  >=65 years | 0 | 2 | 3 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 6
  Male | 5 | 4 | 4 | 5 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 6 | 6 | 5 | 22
  Black or African American | 1 | 0 | 0 | 1 | 2
  Hispanic or Latino | 1 | 2 | 1 | 3 | 7
  Not Hispanic or Latino | 4 | 4 | 5 | 3 | 16
  Ethnicity not reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of PF-07081532
Description: Cmax is the maximum plasma concentration.
Time Frame: At 0 (prior to dose), 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, and 144 hours post dose on Day 1
Population: The PK concentration population included all participants who each received 1 dose of PF-07081532 and in whom at least 1 plasma concentration value was reported. The PK parameter analysis population included all participants who each received 1 dose of PF-07081532 and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Without Hepatic Impairment: Participants without hepatic impairment who received PF-07081532 20mg on Day 1
- Mild Hepatic Impairment: Participants with mild hepatic impairment who received PF-07081532 20mg on Day 1
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment who received PF-07081532 20mg on Day 1
- Severe Hepatic Impairment: Participants with severe hepatic impairment who received PF-07081532 20mg on Day 1
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 2236 (10) | 2121 (18) | 2230 (30) | 1536 (49)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; One-way ANOVA was used on the natural log transformed PK parameters with hepatic function group as a fixed factor. The adjusted mean differences and the corresponding 90% confidence intervals derived from ANOVA were exponentiated to provide estimate of the ratio of adjusted geometric means (Test [hepatic impairment group]/Reference [without hepatic impairment group]) and 90% confidence intervals for the ratio; Test type: Other; ANOVA; Ratio of adjusted geometric means = 94.88, 90% CI 2-sided [70.86 to 127.04] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 99.75, 90% CI 2-sided [74.50 to 133.56] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 68.70, 90% CI 2-sided [51.31 to 91.98] — The ratio and 90% CI are expressed as percentages

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-07081532
Description: AUCinf is the area under the plasma concentration-time profile from time zero extrapolated to infinite time.
Time Frame: At 0 (prior to dose), 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, and 144 hours post dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 43200 (40) | 44010 (61) | 67430 (66) | 41680 (62)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 101.87, 90% CI 2-sided [59.74 to 173.71] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 156.07, 90% CI 2-sided [91.53 to 266.14] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 96.48, 90% CI 2-sided [56.58 to 164.51] — The ratio and 90% CI are expressed as percentages

3. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PF-07081532
Description: AUClast is the area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration.
Time Frame: At 0 (prior to dose), 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, and 144 hours post dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 40990 (39) | 41900 (63) | 62680 (64) | 39800 (63)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 102.21, 90% CI 2-sided [59.91 to 174.39] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 152.91, 90% CI 2-sided [89.62 to 260.90] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 97.08, 90% CI 2-sided [56.90 to 165.65] — The ratio and 90% CI are expressed as percentages

4. Primary Outcome: Fraction of Unbound Drug in Plasma (Fu) of PF-07081532
Description: Fu is the fraction of unbound drug in plasma, which is calculated by Cu/C (where Cu represents unbound concentration and C represents total concentration).
Time Frame: At 0 (prior to dose), 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, and 144 hours post dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Ratio | 0.0002753 (12) | 0.0002568 (38) | 0.0002937 (19) | 0.0006780 (66)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 93.29, 90% CI 2-sided [64.61 to 134.69] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 106.68, 90% CI 2-sided [73.89 to 154.03] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 246.28, 90% CI 2-sided [170.57 to 355.58] — The ratio and 90% CI are expressed as percentages

5. Primary Outcome: Unbound Cmax (Cmax,u) of PF-07081532
Description: Cmax,u is the unbound Cmax.
Time Frame: At 0 (prior to dose), 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, and 144 hours post dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 0.6156 (17) | 0.5448 (42) | 0.6551 (36) | 1.042 (34)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 88.50, 90% CI 2-sided [64.13 to 122.12] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 106.40, 90% CI 2-sided [77.11 to 146.83] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 169.19, 90% CI 2-sided [122.61 to 233.47] — The ratio and 90% CI are expressed as percentages

6. Primary Outcome: Unbound AUCinf (AUCinf,u) of PF-07081532
Description: AUCinf,u is the unbound AUCinf.
Time Frame: At 0 (prior to dose), 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, and 144 hours post dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 11.88 (29) | 11.30 (91) | 19.81 (68) | 28.24 (65)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 95.12, 90% CI 2-sided [52.60 to 172.03] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 166.77, 90% CI 2-sided [92.21 to 301.62] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 237.76, 90% CI 2-sided [131.46 to 430.00] — The ratio and 90% CI are expressed as percentages

7. Primary Outcome: Unbound AUClast (AUClast,u) of PF-07081532
Description: AUClast,u is the unbound AUClast.
Time Frame: At 0 (prior to dose), 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, and 144 hours post dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 11.29 (29) | 10.76 (94) | 18.41 (66) | 27.02 (64)
Statistical Analysis 1: Comparison: Without Hepatic Impairment vs Mild Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 95.34, 90% CI 2-sided [52.67 to 172.59] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 2: Comparison: Without Hepatic Impairment vs Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 163.09, 90% CI 2-sided [90.10 to 295.22] — The ratio and 90% CI are expressed as percentages
Statistical Analysis 3: Comparison: Without Hepatic Impairment vs Severe Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; Ratio of adjusted geometric means = 239.47, 90% CI 2-sided [132.29 to 433.47] — The ratio and 90% CI are expressed as percentages

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE (SAE) was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization/prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; or other serious situations such as important medical events. TEAEs were defined as events that started during the effective duration of treatment (ie, starting on or after the dose of PF-07081532 up to the final follow-up visit). AEs presented below were TEAEs. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE.
Time Frame: Day 1 to Day 36
Population: The safety analysis set included all participants who each took 1 dose of PF-07081532.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  All-causality TEAEs | 1 | 0 | 0 | 1
  Treatment-related TEAEs | 0 | 0 | 0 | 1

9. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Safety laboratory assessments included clinical chemistry, hematology, and urinalysis tests. Number of participants with clinical laboratory abnormalities meeting pre-specified criteria is reported.
Time Frame: From baseline (BL) to Day 7
Population: The safety analysis set included all participants who each took 1 dose of PF-07081532. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Hemoglobin (gram per deciliter [g/dL]) <0.8*lower limit of normal (LLN) | 0 | 0 | 0 | 3
  Hematocrit (%) <0.8*LLN | 0 | 0 | 0 | 2
  Erythrocytes (10^12/liter [L]) <0.8*LLN | 0 | 0 | 0 | 1
  Ery. Mean Corpuscular Volume (femtoliter [fL]) >1.1*ULN | 0 | 0 | 1 | 0
  Ery. Mean Corpuscular Hemoglobin (picogram/cell [pg/cell]) <0.9*LLN | 1 | 0 | 0 | 1
  Platelets (10^9/L) <0.5*LLN | 0 | 0 | 1 | 1
  Neutrophils (10^9/L) <0.8*LLN | 0 | 0 | 0 | 1
  Basophils/Leukocytes (%) >1.2*ULN | 0 | 0 | 1 | 1
  Eosinophils/Leukocytes (%) >1.2*ULN | 0 | 0 | 0 | 2
  Monocytes/Leukocytes (%) >1.2*ULN | 0 | 0 | 0 | 3
  Activated Partial Thromboplastin Time (second [sec]) >1.1*ULN | 2 | 5 | 5 | 5
  Prothrombin Time (sec) >1.1*ULN | 0 | 1 | 2 | 6
  Prothrombin International Normalized Ratio >1.1*ULN | 0 | 1 | 3 | 6
  Bilirubin (milligram per deciliter [mg/dL]) >1.5*ULN | 0 | 0 | 2 | 4
  Direct Bilirubin (mg/dL) >1.5*ULN: number analyzed (Participants) | 0 | 1 | 3 | 4
  Direct Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 2 | 4
  Indirect Bilirubin (mg/dL) >1.5*ULN: number analyzed (Participants) | 0 | 1 | 3 | 4
  Indirect Bilirubin (mg/dL) >1.5*ULN | 0 | 0 | 1 | 3
  Aspartate Aminotransferase (unit per liter [U/L]) >3.0*ULN | 0 | 1 | 0 | 1
  Gamma Glutamyl Transferase (U/L) >3.0*ULN | 0 | 1 | 2 | 1
  Albumin (g/dL) <0.8*LLN | 0 | 0 | 0 | 4
  Urate (mg/dL) >1.2*ULN | 0 | 0 | 1 | 0
  Ketones ≥1 | 0 | 0 | 0 | 2
  URINE Hemoglobin ≥1 | 0 | 0 | 0 | 1
  Urobilinogen ≥1 | 0 | 0 | 1 | 3
  URINE Bilirubin ≥1 | 0 | 0 | 0 | 1
  Leukocyte Esterase ≥1 | 1 | 2 | 1 | 1
  Epithelial Cells (/low-power field [LPF]) ≥6: number analyzed (Participants) | 1 | 2 | 1 | 1
  Epithelial Cells (/low-power field [LPF]) ≥6 | 0 | 0 | 1 | 1

10. Secondary Outcome: Number of Participants With Vital Signs Data Meeting the Pre-defined Categorical Summarization Criteria
Description: Vital signs abnormalities included: seated diastolic blood pressure (BP) increase and decrease from BL of >=20mmHg or absolute value <50mmHg; systolic BP increase and decrease from BL of >=30mmHg or absolute value <90mmHg; pulse rate <40 or >120bpm.
Time Frame: From BL to Day 7
Population: The safety analysis set included all participants who each took 1 dose of PF-07081532.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Diastolic BP Value <50mmHg | 0 | 0 | 1 | 0
  Diastolic BP Increase ≥20mmHg | 1 | 0 | 0 | 1
  Diastolic BP Decrease ≥20mmHg | 0 | 0 | 1 | 0
  Pulse Rate Value <40bpm | 0 | 0 | 0 | 0
  Pulse Rate Value >120bpm | 0 | 0 | 0 | 0
  Systolic BP Value <90mmHg | 0 | 0 | 0 | 0
  Systolic BP Increase ≥30mmHg | 0 | 0 | 0 | 0
  Systolic BP Decrease ≥30mmHg | 0 | 0 | 2 | 0

11. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting the Pre-defined Categorical Summarization Criteria
Description: ECG assessments included PR interval, QT interval, QTcF, and QRS complex. ECG abnormalities included PR interval BL >200msec and max ≥25% increase from BL, or BL ≤200msec and max ≥50% increase from BL, or absolute value ≥300msec; QRS interval percent change from BL ≥50% or absolute value ≥140msec; QTcF change from BL 30- ≤60msec, >60msec, or absolute value 450- ≤480msec, 480- ≤500msec, or >500msec.
Time Frame: From BL to Day 7
Population: The safety analysis set included all participants who each took 1 dose of PF-07081532.
Measure: Count of Participants; unit: Participants
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  PR Interval Value ≥ 300 msec | 0 | 0 | 0 | 0
  PR Interval %Change ≥ 25/50% msec | 0 | 0 | 0 | 0
  QRS Interval Value ≥ 140 msec | 0 | 0 | 0 | 0
  QRS Interval %Change ≥ 50% msec | 0 | 0 | 0 | 0
  QTcF 450 < Value ≤ 480 msec | 0 | 0 | 0 | 3
  QTcF 480 < Value ≤ 500 msec | 0 | 0 | 0 | 0
  QTcF Value > 500 msec | 0 | 0 | 0 | 0
  QTcF 30 < Change ≤ 60 msec | 0 | 0 | 0 | 0
  QTcF Change > 60 msec | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 36
Description: SAEs and nonserious AEs were recorded on the Case Report Form. SAEs were also reported on the Clinical Trial SAE report form to Pfizer Safety within 24h of awareness. Total number at risk below refers to the number of participants evaluable for SAEs/AEs. Unless otherwise noted, all treatment-emergent, all-causality events are reported.
Arm/Group | Without Hepatic Impairment | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Without Hepatic Impairment (N=6) | Mild Hepatic Impairment (N=6) | Moderate Hepatic Impairment (N=6) | Severe Hepatic Impairment (N=6)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT05478603/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT05478603/SAP_001.pdf